CLINICAL TRIAL: NCT00271479
Title: Assay of the Immunogenicity of Fractional Dose Tetravalent A, C, Y, W135 Meningococcal Polysaccharide Vaccine in Africa
Brief Title: Fractional Dose Tetravalent A, C, Y, W135 Meningococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); University of Oslo (Other); Medecins Sans Frontieres, Netherlands (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MB-04-MEN-04
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Last update posted 2006-12-22 (Estimated); Status verified 2006-12

CONDITIONS: Infections, Meningococcal; Meningitis, Meningococcic
Keywords: Meningitis; Dose-Response Relationship, Immunologic; Neisseria meningitidis; Outbreaks; Vaccine; Africa; Uganda; Prevention of Neisseria meningitidis infections; In outbreak contexts in developing countries
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

INTERVENTIONS:
Biological: A, C, Y, W135 meningococcal polysaccharide vaccine

SUMMARY:
Hypothesis:

Lower doses of each A/C/Y/W135 component of the meningococcal polysaccharide vaccine could confer a similar functional immunogenic response as the dose of 50 μg currently being used, and subsequently be equally protective.

The purpose of this study is to evaluate the use of fractional dose tetravalent meningococcal polysaccharide vaccine to control outbreak especially caused by N. meningitidis serogroup W135

Primary Objectives:

* To measure the immunogenicity of a dose corresponding to one fifth of the amount of the licensed meningococcal A/C/Y/W135 polysaccharide vaccine, i.e. 10 μg for each component; and
* To measure the immunogenicity of a dose corresponding to one tenth of the licensed meningococcal A/C/Y/W135 polysaccharide vaccine, i.e. 5 μg for each component.

DETAILED DESCRIPTION:
In 2002, an epidemic of meningococcal disease started in Burkina Faso and Neisseria meningitidis serogroup W135 was identified as the causative organism. This event followed the outbreaks of 2000 and 2001 in Mecca, Saudi Arabia, and was the first large epidemic caused by serogroup W135. Mass vaccination of the population with the only vaccine protecting against W135, i.e. the tetravalent A/C/Y/W135 polysaccharide vaccine (TPSV), was not possible because of the global shortage in supply, in addition to its cost. In 2003, GlaxoSmithKline (GSK) produced a trivalent polysaccharide vaccine A/C/W135 for US$ 1.5. This vaccine was used in Burkina Faso in the new epidemic faced by this country in 2003. However, availability and affordability of the tetravalent A/C/Y/W135 polysaccharide vaccine and of the trivalent A/C/W135 polysaccharide vaccine are still under discussion between the WHO and the producers. The risk of further epidemics due to the W135 strain in other African countries is of high concern for the scientific community.

The current dose of the licensed tetravalent A/C/Y/W135 polysaccharide vaccine contains 50 μg of each polysaccharide component. During the 1980's, researchers from the Walter Reed Army Institute of Research (WRAIR) did extensive works on the immunogenicity of meningococcal polysaccharide vaccines in adults. A first study performed by Griffiss et al. demonstrated that doses of 5 μg of group Y and group W135 polysaccharides were as effective as doses of 50 μg in inducing production of bactericidal antibody amounts correlating with functional immunity (Griffiss et al. Mil Med 1985; 150: 529-33). A second study concluded that doses of 7.5 μg (Y and W) and 15 μg (A and C) were sufficient to induce equivalent binding and bactericidal antibody responses as 50 μg (Griffiss et al. Infect Immun 1982; 37: 205-8). In a more recent study from Granoff et al., 1/50 (1 mcg) of the ordinary dose of tetravalent A/C/Y/W135 vaccine was given (Granoff et al. J Infect Dis 1998; 178: 870-4). The antibody responses to A and C have been measured, and this low dose was sufficient to mount a C response in most of the subjects, but the dose was less effective in eliciting a response to A. The antibody responses to W135 and Y were not reported.

Hypothesis:

Lower doses of each A/C/Y/W135 component of the meningococcal polysaccharide vaccine could confer a similar functional immunogenic response as the dose of 50 μg currently being used, and subsequently be equally protective.

It would potentially bring two major benefits. Firstly, it would increase the number of tetravalent vaccine doses available on the market. Secondly, it would decrease the cost of the individual vaccine dose. As a result, more people could be vaccinated, and thereby protected against the disease, and to a lower price.

Results obtained with the study on the tetravalent A/C/Y/W135 polysaccharide vaccine would be valid for the trivalent A/C/W135 polysaccharide vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers should not be suffering of severe chronic disease or a known congenital or acquired immunodeficiency. A medical exam will be performed by a medical doctor before inclusion.
* Volunteers must be living in the Mbarara district and within 15 km from the site of immunization. Volunteers should be residents of the chosen site and should express no plan of moving from this area during the study period.
* Volunteers must be available for follow-up for the duration of the study (minimum of 24 months).

Exclusion Criteria:

* Volunteers with severe chronic disease or with a general condition requiring hospital admission.
* Volunteers with a known congenital or acquired immunodeficiency (e.g. HIV). Diagnosis will be presumptive based on the medical background and the clinical examination. No serological HIV testing will be performed.
* Evidence of any concomitant infection at the time of presentation (including rashes other than scabies; ear, nose or throat infections; and abnormal respiratory system examination).
* The patient has any other underlying diseases that compromise the diagnosis and the evaluation of the response to the study medication.
* History of serious adverse reactions to vaccines such as anaphylaxis or related symptoms such as hives, respiratory difficulty, angioedema and abdominal pain.
* Malnutrition: The nutritional assessment of children aged 24-59 months, a weight-for-height (W/H) index, will be calculated. This index is expressed in standard deviations of a normalised distribution of a reference population 38 (National Centre for Health Statistics, USA). Children under 5 years old with a Z-score inferior to -2 will be excluded. For children over 5 or adults, the clinical examination will be considered.
* Pregnant women and lactating women are not eligible for this trial. All women of child-bearing age must provide a urine sample for pregnancy testing before inclusion and, for sub-group "b", before the second vaccine injection.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 720
Dates: Start 2004-06; Study Completion 2006-11

PRIMARY OUTCOMES:
To measure the immunogenicity of a dose corresponding to one fifth of the amount of the licensed meningococcal A/C/Y/W135 polysaccharide vaccine, i.e. 10µg for each component
To measure the immunogenicity of a dose corresponding to one tenth of the licensed meningococcal A/C/Y/W135 polysaccharide vaccine, i.e. 5µg for each component

SECONDARY OUTCOMES:
To determine the pharyngeal carriage of N. meningitidis and in particular W135 strains in the study population
To determine the natural immunity towards N. meningitidis serogroup A, C, Y and W135 before immunisation in the study population
To measure a possible waning of immunity at one year and at two years after immunisation
To measure the immune response after challenging with a second dose of the commercialised meningococcal A/C/Y/W135 polysaccharide vaccine after one year, in a group of volunteers who have received a reduced dose on day 0

CONTACTS AND LOCATIONS:
Overall Officials: Philippe J Guerin, MD, MPH, PhD, Principal Investigator — Epicentre; Dominique A Caugant, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (2):
- Norwegian Institute of Public Health, Oslo, Norway
- Mbarara Epicentre Research Base, Mbarara, Uganda

REFERENCES:
- [Background] Griffiss JM, Brandt BL, Broud DD. Human immune response to various doses of group Y and W135 meningococcal polysaccharide vaccines. Infect Immun. 1982 Jul;37(1):205-8. doi: 10.1128/iai.37.1.205-208.1982. PMID 6809627
- [Background] Griffiss JM, Brandt BL, Broud DD, Altieri PL, Berman SL. Relationship of dose to the reactogenicity and immunogenicity of meningococcal polysaccharide vaccines in adults. Mil Med. 1985 Oct;150(10):529-33. No abstract available. PMID 3934585
- [Background] Granoff DM, Gupta RK, Belshe RB, Anderson EL. Induction of immunologic refractoriness in adults by meningococcal C polysaccharide vaccination. J Infect Dis. 1998 Sep;178(3):870-4. doi: 10.1086/515346. PMID 9728562
- [Derived] Guerin PJ, Naess LM, Fogg C, Rosenqvist E, Pinoges L, Bajunirwe F, Nabasumba C, Borrow R, Froholm LO, Ghabri S, Batwala V, Twesigye R, Aaberge IS, Rottingen JA, Piola P, Caugant DA. Immunogenicity of fractional doses of tetravalent a/c/y/w135 meningococcal polysaccharide vaccine: results from a randomized non-inferiority controlled trial in Uganda. PLoS Negl Trop Dis. 2008;2(12):e342. doi: 10.1371/journal.pntd.0000342. Epub 2008 Dec 2. PMID 19048025